CLINICAL TRIAL: NCT06894758
Title: Development of a Rapid Diagnostic Test to Identify Crimean-Congo Haemorrhagic Fever At the Point-of-Care - Research and Development Testing
Brief Title: Development of a Rapid Diagnostic Test to Identify Crimean-Congo Hemorrhagic Fever - Research and Development Testing
Acronym: DETECT-R&D
Status: Not yet recruiting | Type: Observational
Sponsor: Liverpool School of Tropical Medicine (Other)
Collaborators: Ondokuz Mayıs University (Other); Cumhuriyet University (Other)
Responsible Party: Sponsor
Other Study IDs: LSTM 25-017
Record Dates: First submitted 2025-03-12; First posted 2025-03-25 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: Infectious Diseases, Emerging
Keywords: CCHF; Rapid Diagnostic Test; Lateral Flow; RDT; Medical Device
MeSH Terms: conditions — Communicable Diseases, Emerging

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Remnant samples that are suspected of CCHF infection will be stored. This includes both serum and plasma.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- All participants: All participants will suspected of CCHF infection who present at two hospital sites in Türkiye.

SUMMARY:
Background Crimean-Congo Haemorrhagic Fever (CCHF) is a rare disease with a death rate between 10% and 50%, rising to 80% during outbreaks. There are no approved drugs or vaccines, and existing treatments only work if given early. Current diagnosis is slow (2-5 days), delaying treatment, increasing risks, and heightening the chance of other people being infected. The WHO has prioritized developing rapid diagnostic tests (RDTs) to address these issues.

In regions like Afghanistan and Pakistan, delayed diagnosis is especially dangerous, particularly for pregnant women who cannot access emergency care until results are available. To tackle this, the Liverpool School of Tropical Medicine (LSTM) and Global Access Diagnostics (GADx) have created an RDT prototype to detect CCHF viral antigens. Initial testing in Türkiye (2024) showed promising accuracy, meeting WHO's basic standards but further testing is needed to confirm its reliability, especially with fresh samples.

Aims This study will evaluate the RDT using 200 fresh blood and serum samples during the 2025 CCHF season in Türkiye (Sivas and Samsun). If the test meets WHO standards, a clinical trial with 492 patients in CCHF-endemic areas of Türkiye will follow in 2026 to support regulatory approval (CE IVDR and UKCA certification).

Methods Researchers will test 200 fresh samples for diagnostic accuracy and evaluate the impact of storage conditions. This study aims to improve the test's accuracy and stability. Success will advance the development of a fast, reliable diagnostic tool for better CCHF detection and patient care in affected regions.

DETAILED DESCRIPTION:
Background Crimean-Congo Haemorrhagic Fever (CCHF) is a life-threatening disease with a fatality rate ranging from 10% to 50%, and up to 80% in outbreaks. Despite its severity, there are no licensed drugs or vaccines available, and treatment options like Ribavirin are only effective if administered early. The current diagnostic method is slow, taking 2-5 days, which delays treatment, worsens patient outcomes, increases the risk of human-to-human transmission, and strains healthcare resources. Rapid diagnostic tests (RDTs) have been identified as a priority by the WHO to address these challenges.

Delays in diagnosis are particularly critical in regions such as Afghanistan and Pakistan, where suspected CCHF cases, especially among pregnant women, struggle to access emergency care until test results are available. The WHO R&D Blueprint has emphasized the urgent need for point-of-care (POC) tests to reduce diagnosis time and improve patient management.

To meet this need, the Liverpool School of Tropical Medicine (LSTM) and Global Access Diagnostics (GADx) have developed an RDT prototype capable of detecting CCHF viral antigens. This prototype has demonstrated promising sensitivity and specificity, exceeding the WHO's target product profile (TPP) minimum requirements of >80% sensitivity and >90% specificity, with optimal performance defined as >90% sensitivity and >95% specificity. Initial tests in Türkiye in August 2024 showed the prototype achieving sensitivity of 81.2% in 38 prospective samples and 86.4% in 117 retrospective inactivated serum samples, with specificity between 95.5% and 98%.

Further testing in December 2024 with 770 frozen stored samples in Iraq and Türkiye yielded slightly lower performance, potentially due to the effects of freezing and thawing on sample integrity. We hypothesize that freezing alters gene expression, protein stability, and aggregation, impacting test accuracy. Therefore, additional testing with fresh, unfrozen samples is needed to confirm the RDT's reliability before progressing to clinical evaluation.

Aims This study aims to evaluate the RDT using 200 fresh samples collected during the 2025 CCHF season in Sivas and Samsun, Türkiye. If performance aligns with WHO TPP standards, a clinical trial involving 492 patients in CCHF-endemic regions of Türkiye is planned for 2026. The trial data will support regulatory submissions for CE IVDR and UKCA certification.

Methods Before launching the clinical trial, the investigators will conduct further diagnostic accuracy testing on 200 fresh samples (whole blood and serum) to ensure compliance with WHO TPP standards. These samples, pseudonymized and not used for patient management, will also undergo stability testing to assess the impact of storage conditions, including refrigeration for 72 hours (at Sivas site only) and freeze-thaw cycles.

By using optimized RDTs and fresh samples, we aim to improve sensitivity and specificity beyond previous results from December 2024. This study is critical for refining the test, ensuring its effectiveness, and providing essential data on device stability. Ultimately, this research will pave the way for a reliable, rapid diagnostic tool that can significantly enhance CCHF detection and patient outcomes in endemic regions.

ELIGIBILITY:
Inclusion Criteria:

1. Willing to give whole blood samples (in a serum tube and EDTA tube) suspected of CCHF from Türkiye, Department of Infectious Diseases and Clinical Microbiology, Medical Faculty, Sivas Cumhuriyet University, Sivas or the department of Infectious Diseases or Ondokuz Mayis University (OMU) Faculty of Medicine, Department of Clinical Microbiology and Infectious Diseases, Samsun, that have not been frozen or refrigerated.
2. Adults aged 18 or over.

Exclusion Criteria:

None

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants suspected of CCHF infection requiring a standard of care test.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-05 (Estimated); Primary Completion 2025-10 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Diagnostic Accuracy of the RDT | RDT will be performed at the point-of-care and RT-PCR performed 5-7 days after blood draw.
  The principal objective of this study is to evaluate the diagnostic accuracy (novel RDT against RT-PCR) of the RDT using well-characterised fresh whole blood and serum samples from 200 CCHF suspected patients at the point of care.

SECONDARY OUTCOMES:
Sequencing of positive RT-PCR samples | This will be performed near to the end of the study at LSTM in a batch.
  To sequence using MinION (Oxford Nanopore Technologies) for all RT-PCR positive (in at least one of the 3 PCRs selected) below a Ct count of 30. This objective aims to evaluate the sensitivity of the RDT in different CCHF strains.
Survival status of participants | From enrolment to outcome of participant (discharge or death) up to 1 month post presentation
  To obtain survival data on those infected with CCHF, to evaluate the use of the RDT on severe cases.

CONTACTS AND LOCATIONS:
Overall Officials: Ana Cubas Isabel Atienzar, PhD, Principal Investigator — Liverpool School of Tropical Medicine
Locations (2):
- Turkey (Türkiye) (2):
  - Ondokuz Mayis University (OMU) Faculty of Medicine, Department of Clinical Microbiology and Infectious Diseases, Samsun, Samsun
  - Department of Infectious Diseases and Clinical Microbiology, Medical Faculty, Sivas Cumhuriyet University, Sivas, Sivas

IPD SHARING:
Plan to Share IPD: No
This data will be used in conjunction with next years trial for IVDR submission.